CLINICAL TRIAL: NCT03491488
Title: Brain Games: A Crèches-Based Early Intervention Program to Improve Children's Executive Function and Self Control Skills in São Paulo, Brazil
Brief Title: Brain Games to Improve Executive Function in São Paulo, Brazil
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Grand Challenges Canada (Other); Fundação Maria Cecília Souto Vidigal (Unknown); Harvard University (Other); Swiss Tropical & Public Health Institute (Other)
Responsible Party: Principal Investigator, Alexandra Brentani, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1707-09236
Record Dates: First submitted 2018-03-20; First posted 2018-04-09 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Executive Function
Keywords: executive function; Early childhood education; self regulation
MeSH Terms: conditions — Self-Control

STUDY DESIGN:
Intervention Model Description: randomized controlled trial at 60 public crèches in São Paulo, Brazil
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): 300 children in the randomly selected crèche classrooms receiving the Brain Games intervention.
  The Brain Games intervention we propose in this project is designed to complement and improve current government efforts. Given the importance of executive functioning skills and the high plasticity around age three, early programs like the ones proposed here may be the most effective tool to reduce socioeconomic and intergenerational disparities, and thus nicely complement current social protection policies.
  Interventions: Other: Brain Games
- Control Group (No Intervention): 300 children in the randomly selected creches classrooms receiving the regular Brazilian curriculum.

INTERVENTIONS:
Other: Brain Games — The Brain Games intervention package is used as a tool to improve children's self-regulation and executive function skills. Brain Games were developed as part of larger behavioral intervention package in the US, and are designed to build the fundamental self-regulation skills that children need to be successful in school as well as later in life. The games are designed to be played in the classroom between regular activities.
  Arms: Intervention Group

SUMMARY:
A growing body of research has highlighted the critical importance of children's self-regulation and executive function skills for their school performance as well as for their later life outcomes. Starting around age three, children have a unique potential to improve these skills and establish positive behaviors that will support them in school and life.

This project will adapt, implement and evaluate the effectiveness of the Brain Games intervention package as a tool to improve children's self-regulation and executive function skills. Brain Games were developed as part of larger behavioral intervention package in the US, and are designed to build the fundamental self-regulation skills that children need to be successful in school as well as later in life. The Brain Games curriculum will be adapted to Brazil, and evaluated through a 12 month randomized controlled trial with 60 crèches in São Paulo to assess its impact on children's self-regulation and executive functioning skills.

DETAILED DESCRIPTION:
Even though Brazil has made major efforts to improve children's access to early childhood care and education, most of Brazil's (as well as other countries') early childhood programming focuses on care and early learning including early literacy and numeracy. Relatively little attention is currently given to the development of the non-academic self-regulation and executive function skills that have been shown to be critical for children's schooling as well as later life outcomes. The main idea of this project is to adapt Brain Games - an evidence-based, scalable intervention package developed for the US - to the Brazilian context, and to assess its impact on children's self-regulation and executive functioning skills through a randomized controlled trial.

The Brain Games package consists of a series of games and exercises designed for young children in classroom settings. Brain Games are a new, "kernelized" approach to intervention, with simple and discrete stand-alone activities that can be easily integrated into routine operations at crèches with a limited amount of training and supervision of center staff.

The proposed project embodies the principle of Integrated Innovation; the main scientific innovation is the development and validation of a new, kernelized executive functioning intervention package for Brazil. The intervention package will be designed for, and implemented through the public early childhood care section; from a social perspective, the main innovation is to increase the quality of care socially disadvantaged children obtained in public child care. From a business perspective, the intervention itself is sustainable and scalable, as its main elements have already been developed in the US, training is minimal, and material costs are low. Furthermore, the intervention consists of games that are easy and fun to play for children, and can be easily added to the existing curriculum. If the trial is successful, the intervention package could and likely would be rolled out at larger scale.

ELIGIBILITY:
Inclusion Criteria:

* age 3 years, 0 days to 4 years, 364 days at baseline
* attending public creches and pre-schools São Paulo's Western region

Exclusion Criteria:

* children younger than 3 years or older than 4 years at baseline
* not attending public creches and pre-schools

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2018-04-16 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Child executive functions | Endline assessements - after 12 months of intervention delivery, scheduled for April 2019
  Child executive functions will be a composite score based on three tests conducted with all children at endline: a hearts-and-flowers test conducted on tablets, a pencil-tap test, and the IDELA executive functioning assessment. The composite score will be computed using principal component analysis of the normalized scores in the three tests.

SECONDARY OUTCOMES:
School readiness | Endline survey - after 12 months of intervention; scheduled for April 2019
  School readiness will be assessed using the IDELA tool

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Brentani, PhD, Principal Investigator — USao Paulo
Locations (1):
- Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Intervention materials will be shared with the Government.